CLINICAL TRIAL: NCT02933749
Title: Effects of the Prone and the Sitting Positions on the Brain Oxygenation in Posterior Fossa Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Özlem Korkmaz Dilmen, MD, DESA, Associate Prof in Anesthesiology, Istanbul University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: Istanbul
Record Dates: First submitted 2016-10-10; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Infratentorial Neoplasms
MeSH Terms: conditions — Infratentorial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The sitting (Active Comparator): The sitting position Device sCtO2 Device BIS
  Interventions: Device: SctO2; Device: BIS
- The prone (Active Comparator): The prone position Device sCtO2 Device BIS
  Interventions: Device: SctO2; Device: BIS

INTERVENTIONS:
Device: SctO2 — The non invasive cerebral oxymetry (INVOS-Covidien) has been used to measure cerebral oxygen saturation.
  Other Names: INVOS-Covidien
Device: BIS — Bispectral index

SUMMARY:
The sitting or prone positions are used for posterior fossa surgery. Although the sitting position may cause hemodynamic instability, venous air embolism, it also provides optimum access to midline lesions, decreases intracranial pressure. The sitting position has not been only used in neurosurgery, it has been also used in the shoulder surgery. The sitting position related hypotension may reduce the cerebral perfusion pressure, therefore may cause cerebral ischemia. The sitting position related cerebral ischemia has been shown in the shoulder surgery. The non invasive cerebral oxymetry (INVOS-Covidien) has been used to measure cerebral oxygen saturation. Some studies has been done to investigate whether the sitting position cause cerebral desaturation or not in the shoulder surgery by non invasive cerebral oxymetry. The study results are controversial.

It has been investigated that the effect of the prone position on the cerebral oxygenation in the spine surgery and the investigators found that the prone position may increase cerebral oxygenation.

However, all studies have been done in patients without intracranial pathology. We speculate that due to the sitting position reduces the intracranial pressure, it may improve the cerebral oxygenation in the patients have intracranial pathology. Therefore we will compare the sitting and the prone positions effects on the cerebral oxygenation in patients undergoing posterior fossa tumour surgery by non invasive cerebral oxymetry.

Method: 62 patients have posterior fossa tumour will include the study. Patients will divide to 2 groups according to the surgical position, the prone (n=31) or the sitting (n=31). Patients heart rate, mean blood pressure (MAP), cerebral oxygen saturation (SctO2), peripheral oxygen saturation (SpO2), BIS values will record before the induction of anesthesia. Five minutes after the standard anesthesia induction all values will record and it will accept as a baseline. After that all these parameters will record in each 3 minutes until the beginning of surgery. Mean while, more than 5 % reduction in SctO2 and more than 20 % reduction in SctO2 and/or MAP will record. As well as, if the SctO2 reduces than 55 and 60 %, it will record.

DETAILED DESCRIPTION:
The sitting or prone positions are used for posterior fossa surgery. Although the sitting position may cause significant complications such as including hemodynamic instability, venous air embolism, paradoxical air embolism (PAE), pneumocephalus, peripheral neuropathy, quadriplegia and macroglossia, it also provides optimum access to midline lesions in posterior fossa and cervical spine, improves blood and cerebral spinal fluid drainage, decreases intracranial pressure, lowers airway pressure, and improves access to the endotracheal tube and ability to observe the face for signs of cranial nerves stimulations. The sitting position has not been only used in neurosurgery, it has been also used in the shoulder surgery. The sitting position related hypotension may reduce the cerebral perfusion pressure, therefore may cause cerebral ischemia. The sitting position related cerebral ischemia has been shown in the shoulder surgery.

The non invasive cerebral oxymetry (INVOS-Covidien) has been used to measure cerebral oxygen saturation. Some studies has been done to investigate whether the sitting position cause cerebral desaturation or not in the shoulder surgery by non invasive cerebral oxymetry. The study results are controversial.

It has been investigated that the effect of the prone position on the cerebral oxygenation in the spine surgery and the investigators found that the prone position may increase cerebral oxygenation.

However, all studies have been done in patients without intracranial pathology. We speculate that due to the sitting position reduces the intracranial pressure, it may improve the cerebral oxygenation in the patients have intracranial pathology. Therefore we will compare the sitting and the prone positions effects on the cerebral oxygenation in patients undergoing posterior fossa tumour surgery by non invasive cerebral oxymetry.

Method: 62 patients have posterior fossa tumour will include the study. Patients will divide to 2 groups according to the surgical position, the prone (n=31) or the sitting (n=31). Patients heart rate, mean blood pressure (MAP), cerebral oxygen saturation (SctO2), peripheral oxygen saturation (SpO2), BIS values will record before the induction of anesthesia. Five minutes after the standard anesthesia induction all values will record and it will accept as a baseline. After that all these parameters will record in each 3 minutes until the beginning of surgery. Mean while, more than 5 % reduction in SctO2 and more than 20 % reduction in SctO2 and/or MAP will record. As well as, if the SctO2 reduces than 55 and 60 %, it will record.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infratentoril neoplasms

Exclusion Criteria: Stroke

* Diabetes mellitus
* Chronic obstructive pulmonary disease
* Anemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Cerebral oxygen saturation | Change from baseline cerebral oxygen saturation up to skin incision
  After anesthesia induction cerebral oxygen saturation will record in each 3 minutes until the beginning of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Korkmaz Dilmen, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Ozlem Korkmaz Dilmen, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Dilmen OK, Akcil EF, Tureci E, Tunali Y, Bahar M, Tanriverdi T, Aydin S, Yentur E. Neurosurgery in the sitting position: retrospective analysis of 692 adult and pediatric cases. Turk Neurosurg. 2011;21(4):634-40. PMID 22194128
- [Background] Pohl A, Cullen DJ. Cerebral ischemia during shoulder surgery in the upright position: a case series. J Clin Anesth. 2005 Sep;17(6):463-9. doi: 10.1016/j.jclinane.2004.09.012. PMID 16171668
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS, Vaughn J, Nisman M. Cerebral oxygen desaturation events assessed by near-infrared spectroscopy during shoulder arthroscopy in the beach chair and lateral decubitus positions. Anesth Analg. 2010 Aug;111(2):496-505. doi: 10.1213/ANE.0b013e3181e33bd9. Epub 2010 May 27. PMID 20508134